CLINICAL TRIAL: NCT04715438
Title: Vaccination Against cOvid In CancEr
Brief Title: Vaccination Against COVID-19 in Cancer
Acronym: VOICE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202000865
Record Dates: First submitted 2021-01-11; First posted 2021-01-20 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: vaccination; COVID-19; solid tumors; immune response
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A: Individuals without cancer (Experimental): A cohort of individuals without a cancer diagnosis is included for comparison. Because age is an important predictor of the ability to mount an effective immune response to vaccination, partners of patients in cohort B, C, and D.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine from Moderna
- Cohort B: patients receiving immunotherapy (Experimental): Cancer patients receiving immunotherapy
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine from Moderna
- Cohort C: patients receiving chemotherapy (Experimental): Cancer patients receiving chemotherapy
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine from Moderna
- Cohort D: patients receiving chemo-immunotherapy (Experimental): Cancer patients receiving chemo-immunotherapy
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine from Moderna

INTERVENTIONS:
Biological: mRNA-1273 SARS-CoV-2 vaccine from Moderna — All participants will receive two vaccinations against COVID-19 according to standard of care.

SUMMARY:
This study will collect information on immune response and adverse events after vaccination against coronavirus disease (COVID-19) in a vulnerable patient cohort. Understanding the ability or disability to mount a protective immune response after vaccination will help to counsel patients during the pandemic and support decisions on whom to vaccinate and to identify patients who require other measures to protect them from COVID-19.

DETAILED DESCRIPTION:
Rationale:

Patients with cancer have an increased risk of adverse outcome of COVID-19, which is determined by their underlying disease and/or cancer treatment. Therefore, vaccination of cancer patients against COVID-19 is recommended. However, phase III studies do not provide robust information on efficacy and safety in this vulnerable population. In patients with cancer, the disease itself, but also immunotherapy and chemotherapy, may have a significant impact on the ability to develop an effective immune response to COVID-19 vaccination, and could even increase the risk of adverse events.

Objective:

To assess immune response and adverse events after administration of one approved vaccine against COVID-19 in patients with cancer treated with immunotherapy and/or chemotherapy.

Study design:

This is a prospective multicenter, multicohort study.

Study population:

Four cohorts will receive vaccination against COVID-19:

A. Individuals without cancer (N=246, i.e., partners of patients in cohort B, C, and D) B. Patients with cancer treated with immunotherapy (N=135) C. Patients with cancer treated with chemotherapy (N=246) D. Patients with cancer treated with chemo-immunotherapy (N=246)

Intervention:

Participants will be vaccinated against COVID-19 with an approved vaccine. Blood will be drawn at different time points by venipuncture and mucosal lining fluid will be collected at 2 time points.

Main study parameters/endpoints:

The primary endpoint is the antibody based immune response on day 28 after the second vaccination. Participants will be classified as responders or non-responders. The definition of response is seroconversion defined as presence of SARS-CoV-2 spike S1-specific IgG antibodies in individuals without measurable anti-S antibodies at baseline. Participants who are seropositive at baseline will not be included in the analysis of the primary endpoint. The percentage of responders of each patient cohort will be compared with the percentage responders in the control group. Safety is a secondary endpoint which will be reported in terms of percentage of solicited local and systemic adverse events (AEs) graded according to severity. Other secondary endpoints include longevity at 6 months and levels of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) specific T cell responses.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Participants will have to visit the hospital at 6 time points and participants who receive a third vaccination will have 2 additional hospital visits. The vaccine will be administered two times according to standard of care, with the option of a third vaccination for participants without an adequate response after 2 vaccinations. Blood will be drawn (~373 ml in total for participants receiving 2 vaccinations, and ~539ml in participants receiving 3 vaccinations) prior to the vaccinations and at day 28 and 6 months, 11 months and 18 months after the second vaccination. Nasal mucosal lining fluid samples will be collected at baseline and day 28 after the second vaccination in a subgroup of patients. Blood sampling will give minor discomfort. Vaccination can cause AEs including fatigue, chills, headache, myalgia, and pain at the injection site. For seven days after each vaccination, participants will be asked to record local and systemic reactions using a questionnaire. At baseline and at 3, 6, 9, 12, 15 and 18 months after the second vaccination, patients will be asked to complete questionnaires about potential subsequent testing for SARS-CoV-2, diagnosis of COVID-19, and severity of COVID-19.

This study will collect information on immune response and adverse events after vaccination against COVID-19 in a vulnerable patient cohort. It will also explore immune response and safety of a third vaccination in participants without an adequate antibody response after the second vaccination. Understanding the ability or disability to mount a protective immune response after vaccination will help to counsel patients during the pandemic and support decisions on whom to vaccinate and to identify patients who require other measures to protect them from COVID-19. Participants will be informed about their antibody titer in a letter that includes an explanation about what this means to them. This will be done after antibody measurements have been completed for day 28 after second vaccination, and again after completion of measurements for 6 months and 28 days after third vaccination, and 11 months and 18 months after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, a subject must meet all of the following criteria:

* Age of 18 years or older
* Life expectancy > 12 months
* Ability to provide informed consent

Additional criteria for cohort A:

• Partner of a participating patient

Additional criteria for cohort B:

* Histological diagnosis of a solid malignancy
* Treatment with monotherapy immune checkpoint inhibitor (ICI) against Programmed Death 1 (PD1) or its ligand PD-L1 (in curative or non-curative setting)
* Last ICI administration within 3 months of vaccination

Additional criteria for cohort C:

* Histological diagnosis of a solid malignancy
* Treatment with cytotoxic chemotherapy (monotherapy and combination chemotherapy is allowed, as well as a combination with radiotherapy, in curative or non-curative setting)
* Last chemotherapy administration within 4 weeks of vaccination

Additional criteria for cohort D:

* Histological diagnosis of a solid malignancy
* Treatment with a PD1 or PD-L1 antibody in combination with cytotoxic chemotherapy (in curative or non-curative setting)
* Last chemotherapy administration within 4 weeks of vaccination
* Last ICI administration within 3 months of vaccination

Exclusion criteria:

* Confirmed SARS-CoV-2 infection (current or previous)
* Women who are pregnant or breastfeeding
* Active hematologic malignancy
* Any immune deficiency not related to cancer or cancer treatment (e.g. inherited immune deficiency or known infection with Human Immunodeficiency Virus)
* Systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medication within 14 days of vaccination. Inhaled or topical steroids, and adrenal replacement steroids (> 10 mg daily prednisone equivalent) are permitted. In addition, standard of care with short course steroids to prevent nausea and allergic reactions from chemotherapy or iodinated CT contrast is allowed.

Additional criteria for cohort A:

* Current or previous diagnosis of a solid malignancy, unless treated with curative intent >5 years before enrolment and without signs of recurrence during proper follow-up
* Previous history of a hematologic malignancy

Additional criteria for cohort B:

• Treatment with cytotoxic chemotherapy within 4 weeks of vaccination

Additional criteria for cohort C:

• Treatment with an ICI within 3 months of vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 791 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Immune response to vaccination against COVID-19 measured as antibody response expressed as geometric mean concentration: arbitrary units (AU)/ml | Measured at 28 days after vaccination
  The primary endpoint is the antibody based immune response to vaccination against COVID-19 on day 28 after the second vaccination in patients receiving cancer treatment as compared to individuals without cancer. Expressed as antibody response expressed as geometric mean concentration: arbitrary units (AU)/ml

SECONDARY OUTCOMES:
Safety assessment (S)AEs; Incidence and severity of solicited AEs during 7 days after each vaccination with incidence and nature of SAEs reported during 7 days after each vaccination | During 7 days after vaccination
  * Incidence and severity of solicited AEs during 7 days after each vaccination
  * Incidence and nature of SAEs during 7 days after each vaccination
Safety assessment immune related (ir), with incidence and nature of newly occurring irAEs grade ≥ 3 in cohort B and D reported up to 28 days | From start till 28 days after second vaccination
  - Incidence and nature of newly occurring irAEs grade ≥ 3 in cohort B and D up to 28 days after the last vaccination graded according to the Common Criteria for Adverse Events version 5.0 (CTCAE v5.0)
  * Neutralizing capacity of antibodies to test functionality
  * Assessment of SARS-CoV2 specific T cells response, 7 days, 28 days, and 6 months after vaccination using a high throughput Interferon ɣ ELIspot.
Safety assessment AE of special interest (SI)s with Incidence, nature and severity of AESIs graded according to CTCAE v5.0 reported up to 12 months after vaccination | From start till 12 months after vaccination
  - Incidence, nature and severity of AESIs graded according to CTCAE v5.0
Assessment of immune response: expressed as geometric mean antibody concentration: arbitrary units (AU)/ml | measured at 6 to 18 months after vaccination
  Persistence of antibody response expressed as geometric mean concentration: arbitrary units (AU)/ml
Assessment of immune response: measured as levels of SARS-CoV-2 specific T-cell responses expressed as number of IFNg producing T cells/ million peripheral blood mononuclear cells (PBMCs) | measured 28 days to 18 months after vaccination
  Levels of SARS-CoV-2 specific T-cell responses expressed as number of IFNg producing T cells/ million peripheral blood mononuclear cells (PBMCs)

CONTACTS AND LOCATIONS:
Overall Officials: E G de Vries, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (3):
- Netherlands (3):
  - NKI-AvL, Amsterdam
  - UMCG, Groningen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
Alignment and reuse Our options for reusing data, biological materials, and/or other resources (from research or practice) in your project.
  * Data: Clinicopathological parameters as described in the protocol
  * Biological materials: Blood
  * Research software: R statistical package, Castor, MOLGENIS
  * Other resources, i.e.,Nederlandse Kankerregistratie (NKR), the Dutch Cancer Registry, electronic patient dossiers (EPDs)
  FAIR data within the COVID-19 research community
  * A COVID-19 related or other Findability, Accessibility, Interoperability, and Reuse (FAIR) data points
  * COVID-19 research platform for data sharing
  we will make protocol etc. available on the website soon voicetrial.nl
Supporting Information: Study Protocol
Time Frame: we start the make interim results available second half of 2021
Access Criteria: we aim to share as much as possible also through own website, and COVID-19 platforms that are considered for this kind of research

REFERENCES:
- [Derived] Piening A, Ebert E, Khojandi N, Alspach E, Teague RM. Immune responses to SARS-CoV-2 in vaccinated patients receiving checkpoint blockade immunotherapy for cancer. Front Immunol. 2022 Dec 13;13:1022732. doi: 10.3389/fimmu.2022.1022732. eCollection 2022. PMID 36582225
- [Derived] Oosting SF, van der Veldt AAM, GeurtsvanKessel CH, Fehrmann RSN, van Binnendijk RS, Dingemans AC, Smit EF, Hiltermann TJN, den Hartog G, Jalving M, Westphal TT, Bhattacharya A, van der Heiden M, Rimmelzwaan GF, Kvistborg P, Blank CU, Koopmans MPG, Huckriede ALW, van Els CACM, Rots NY, van Baarle D, Haanen JBAG, de Vries EGE. mRNA-1273 COVID-19 vaccination in patients receiving chemotherapy, immunotherapy, or chemoimmunotherapy for solid tumours: a prospective, multicentre, non-inferiority trial. Lancet Oncol. 2021 Dec;22(12):1681-1691. doi: 10.1016/S1470-2045(21)00574-X. Epub 2021 Nov 9. PMID 34767759

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT04715438/Prot_SAP_002.pdf